CLINICAL TRIAL: NCT01434797
Title: Prospective Study on the Usefulness and Diagnostic Value of F-18-FDG PET/CT in the Diagnosis of Permanent Central Venous Catheters Infection
Brief Title: Value of PET/CT Imaging in the Diagnosis of Permanent Central Venous Catheters Infection
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, John O. Prior, Centre Hospitalier Universitaire Vaudois, Nuclear Medicine, University of Lausanne Hospitals
Other Study IDs: 89/11
Record Dates: First submitted 2011-09-01; First posted 2011-09-15 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Infection
Keywords: Infection; Permanent central venous catheter; Device Related
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Confirmed CVCP infection before removal: Patients with permanent central venous catheter infection confirmed by conventional method
- Presumed CPVP infection before removal: Patients with probable permanent central venous catheter infection (standard methods for infection detection not conclusive)
- Uninfected CVCP before removal: Patients with planned permanent central venous catheter removal (no infection)

SUMMARY:
The study hypothesis is that F-18-FDG PET/CT and microcalorimetry might have a diagnostic value in the detection of permanent central venous catheters (PCVC) infection when conventional means of PCVC infection detection are non-conclusive.

DETAILED DESCRIPTION:
Permanent central venous catheters are frequently infected and therefore need surgical removal. When a clear diagnostic for infection cannot be defined, catheter removal might be at risk for the patient, for the therapeutic follow-up and in terms of costs. PET/CT and microcalorimetry might help giving conclusive diagnostic of catheter infection.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed catheter infection requiring surgical removal
* patients with probable catheter infection requiring surgical removal
* patients with planned removal of uninfected catheter
* ≥18years old

Exclusion Criteria:

* extreme claustrophobia
* pregnancy and breastfeeding
* severe septicemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathology requiring permanent central venous catheter will be selected mainly from nephrology and oncology departments . They might also be selected from other deparments.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic value (sensitivity and sensibility, positive/negative predictive value) of F-18-FDG PET/CT imaging in the detection of CVCP infection | 6 months
  To determine the clinical use of PET/CT in the detection of catheter infection by comparing PET/CT imaging results to standard means of catheter infection detection (i.e. clinical signs and hemoculture [positive or negative])

SECONDARY OUTCOMES:
Diagnostic value (sensitivity and sensibility, positive/negative predictive value) of microcalorimetry in the detection of CVCP infection | 6 months
  To determine the clinical use of microcalorimetry in the detection of catheter infection by comparing microcalorimetry results to standard means of catheter infection detection (i.e. clinical signs and hemoculture [positive or negative])

CONTACTS AND LOCATIONS:
Overall Officials: John O Prior, PhD MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois and University of Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Nuclear Medicine, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No